CLINICAL TRIAL: NCT07085988
Title: Nutritional Management During Concurrent Chemoradiotherapy for Nasopharyngeal Carcinoma Has an Impact on Immunonutritional Status and Therapeutic Phase Toxicity and Prognostic Effects
Brief Title: Effect of Nutritional Management on Patients With Concurrent Chemoradiotherapy for Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangxi Provincial Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Jiangxi Cancer Hospital
Record Dates: First submitted 2025-04-07; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Nasopharyngeal Carcinoma (NPC)
Keywords: Nasopharyngeal Carcinoma; Concurrent chemoradiotherapy; Immunonutrition Lymphocyte count
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Effect of nutritional management in patients with nasopharyngeal carcinoma (Experimental): Patients with nasopharyngeal carcinoma are given rapid gamin during concurrent chemoradiotherapy
  Interventions: Other: Rapid glitter

INTERVENTIONS:
Other: Rapid glitter — Patients with nasopharyngeal carcinoma are given rapid gamin during concurrent chemoradiotherapy

SUMMARY:
Nasopharyngeal carcinoma (NPC) is a malignant tumor that develops in the nasopharyngeal mucosal epithelium. Due to the disease itself and the impact of anti-tumor therapy, malnutrition has become a common clinical complication in patients with NPC, among which NPC patients receiving concurrent chemoradiotherapy are one of the groups with the highest incidence of malnutrition, and malnutrition seriously affects the prognosis of NPC patients. Nutritional management throughout the course has a positive impact on the prognosis and life management of NPC patients. As an immune-enhancing oral nutritional preparation, it is helpful to maintain the weight and immune function of patients with nasopharyngeal carcinoma during concurrent chemoradiotherapy, reduce the degree of treatment-related side effects during concurrent chemoradiotherapy for nasopharyngeal carcinoma, and delay the occurrence of acute side effects. The purpose of this study was to investigate the effect of rapid rapid rapid improvement of patients' immune status during concurrent chemoradiotherapy, and to further evaluate its impact on patients' weight, prognosis, treatment-related toxic side effects, and quality of life. In this study, 109 patients with nasopharyngeal carcinoma who received concurrent chemoradiotherapy in our hospital are planned to be included, and all patients in this group will be given oral tachyphin at a standard dose from the first day of radiotherapy. The nutritional immune status of the patient was assessed at different points during the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* 1.Patients with nasopharyngeal carcinoma confirmed by histopathology;2.Clinical stage stage II-IVa,Concurrent chemoradiotherapy is included in the definitive treatment regimen;3.Age ≥ 18 years, male or female;4.PG-SGA score of 0-8 before radiotherapy;5.KPS score ≥ 60 or ECOG score ≤3;6.Nutritional supplementation can be given by mouth or enterally;7.Patients sign a formal informed consent form to indicate that they understand that this study complies with hospital policies;8.Serum hemoglobin ≥ 90 g/L, platelet ≥ 100×109/L, absolute neutrophil count ≥ 1.5×109/L;9.serum creatinine ≤1.25 times ULN or creatinine clearance ≥60 mL/min;10.Serum bilirubin ≤ 1.5-fold ULN, AST (SGOT) and ALT (SGPT) ≤ 2.5-fold ULN, and alkaline phosphatase ≤ 5-fold ULN.

Exclusion Criteria:

* 1.Have a second primary tumor;2.Those who do not receive concurrent chemoradiotherapy;3.Comorbid diabetes mellitus, or history of severe endocrine and metabolic diseases;4.Those who are allergic to oral nutritional meal replacements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Decreased proportion of immune cell subsets | 2 weeks
  The proportion of immune cell subsets that decline during chemoradiotherapy, including CD3, CD4, CD8

SECONDARY OUTCOMES:
Change in the patient's weight | 2 weeks
  Change in the patient's weight during concurrent chemoradiotherapy
Disease Free Survival | 3 Years
  DFS was defined as the interval from the date of diagnosis to the data of disease recurrence or death DFS was defined as the interval from the date of diagnosis to the data of disease recurrence or death DFS was defined as the interval from the date of diagnosis to the data of disease recurrence or death

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangxi Cancer Hospital, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No